CLINICAL TRIAL: NCT06355284
Title: Pathways to Hope: Pilot fMRI Study of OCPD and Suicide Risk in Trauma-Exposed Veterans
Brief Title: Overcontrol and Suicide in PTSD
Acronym: OSP
Status: Recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: D5150-P
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Compulsive Personality Disorder; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Compulsive Personality Disorder; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: None Retained — No biospecimens retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Overcontrol: Trauma-exposed veterans with PTSD symptoms and average rigidity, emotional overcontrol, and maladaptive perfectionism subscale scores on the Pathological Obsessive Compulsive Personality Scale greater than or equal to 4.
  Interventions: Other: Functional MRI

INTERVENTIONS:
Other: Functional MRI — While in the MRI scanner, participants will complete several classic experimental tasks designed to capture brain activity related to core cognitive features of overcontrol that impact social functioning. Tasks include the Stop Signal Task (error monitoring), Delay Discounting Task (valuation, impulsivity), and Reversal Learning (cognitive flexibility).

SUMMARY:
High standards and self-discipline are prized in military culture, but drawbacks of overcontrol are often ignored. Overcontrol is characterized by over-regulated behavior and cognitive rigidity, driven by an intense need for perfection and control. It is frequently observed in people with obsessive-compulsive (OC) spectrum disorders, especially OC Personality Disorder (OCPD). Their inclination to set high expectations for others can strain social bonds. When grappling with mental health challenges, overcontrolled individuals often do so with limited social support, and as a result, tend to be at greater risk of developing more severe mental health symptoms, or suicidal thoughts and behaviors, over time.

New treatments are needed to improve social functioning in these vulnerable Veterans. Adding brain stimulation to psychotherapy is one method that might speed learning of social skills discussed in therapy. However, before this technology can be developed and tested more broadly, the investigators must make sure that the methods used to measure social functioning and related brain circuits are acceptable to most potential patients and can be used consistently.

In this pilot project, the investigators aim to recruit trauma-exposed Veterans with overcontrolled traits and study the feasibility and acceptability of:

1. Our recruitment strategy and social functioning and mental health symptom assessments
2. A three-session, weekly fMRI protocol.
3. A three-week online protocol for remote monitoring of social and emotional functioning.

DETAILED DESCRIPTION:
High standards and self-discipline are prized in military culture, but drawbacks of overcontrol are often ignored. Overcontrol, a transdiagnostic phenotype, is characterized by over-regulated behavior and cognitive rigidity, driven by an intense need for perfection and control. It is prevalent in obsessive-compulsive (OC) spectrum disorders, especially OC Personality Disorder (OCPD). Their inclination to set high expectations for others often causes interpersonal tension straining social bonds. When grappling with mental health challenges, overcontrolled individuals often do so with limited social support and consequently, may have poorer outcomes.

Treatments enhancements are needed to improve interpersonal functioning, quality of life and mitigate suicide risk these vulnerable Veterans. Neuromodulation adjunctive to psychotherapy is a promising option. Key obstacles, however, impede the development of circuit-based treatments tailored to this phenotype: 1) limited validation of existing associations between interpersonal functioning and OCPD in a broader, overcontrolled sample, 2) the absence of a unified, transdiagnostic circuit model of overcontrol, and 3) robust methods for tracking gradual changes in individuals' functioning throughout the course of treatment.

This pilot project will develop methods to address these knowledge gaps. Specifically, the investigators aim to:

1. Assess the feasibility of our recruitment strategy and evaluate interpersonal functioning in a cohort of trauma-exposed Veterans exhibiting overcontrolled traits.
2. Test the feasibility and acceptability of a three-session, weekly fMRI protocol focused on the circuitry of overcontrol, while evaluating within-subject reliability of observed neural correlates.
3. Examine the feasibility and acceptability of a three-week protocol for remote monitoring of weekly variance in socio-occupational functioning and emotional regulation.

In service of these Aims, the investigators plan to enroll and screen up to 74 Veterans aged 18-65 who are currently receiving care at either PVAMC's Trauma Recovery Clinic (TRC) or Women's Health Clinic (WHC), the latter included to boost female participation. All those who consent to participate will complete the screening assessment. Of these 74 screened participants, the investigators anticipate that 36 Veterans will meet our inclusion/exclusion criteria and will be invited to complete additional psychosocial assessments. A subset of participants (up to n=18) will be invited to complete three MRI sessions and six brief at-home assessments asking questions about stress, emotional regulation, and socio-occupational functioning.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion:

* All prospective participants must be able to comprehend the study's procedures and associated risks and be capable of providing informed consent.
* Mean scores on at least three subscales of the Pathological Obsessive Compulsive Personality Scale (POPS) must be greater than an average score of four (4 = "slightly agree") across subscale items.

  * The POPS is a 49-item self-report assessment of maladaptive behaviors and thought patterns associated with OCPD.
* While Veterans with primary psychotic disorders will be excluded, the presence of other disorders related to obsessive-compulsive tendencies or personality will not be grounds for exclusion.
* Psychiatric medication usage will be assessed during enrollment, but this will not serve as an inclusion or exclusion criterion (with an additional stipulation outlined below for the MRI subsample).

Exclusion Criteria:

General Exclusion:

* The Mini International Neuropsychiatric Interview (M.I.N.I.) will be used to exclude participants with current psychosis or with past psychosis that was unrelated to depression.

Additional MRI Criteria:

* Participants interested in taking part in the MRI portion of the study will undergo a thorough screening to ensure MRI compatibility (e.g., absence of metal in the body, absence of claustrophobia).
* Interested participants must meet the following additional criteria:

  * no medical contraindications for MRI (e.g., pacemakers, non-MRI safe implanted devices)
  * absence of neurological disorders
  * no moderate-to-severe traumatic brain injury (e.g., head trauma with loss of consciousness >5 minutes)
  * no ongoing poorly controlled substance use disorder.
* Lifetime history of seizures, primary or secondary CNS tumors, stroke, or cerebral aneurysm will also be exclusionary.
* For participants in the MRI segment of the study, continued medication use will not be a disqualifying factor if the medication regimen has remained stable for the past month, with no intentions of altering dosages during the study duration.
* This medication criterion will not be applied to participants who do not complete MRI scans.
* For this feasibility trial, individuals exhibiting active suicidal behavior or a score >3 on the suicidal ideation module of the Columbia-Suicide Severity Rating Scale will be ineligible.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include Veterans 18-65 years old. They will be men or women from the greater Providence area receiving care at the VA who have been discharged from active duty, or who served in the National Guard or reserve units. Over 15 months, the investigators plan to screen 74 Veterans aged 18-65 receiving care in VAPHS's Trauma Recovery Clinic (TRC) and Women's Health Clinic (WHC), the latter included to boost female participation.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of potential participants screened per month meeting the overcontrol criterion. | 18 months
  Indexes feasibility of recruitment and enrollment screening strategy.
Percentage of sessions completed by participants receiving MRI. | 22 months
  Indexes feasibility of functional MRI protocol.
Percentage of remote questionnaires completed. | 22 months
  Indexes feasibility of remote measurement of socio-occupational functioning and emotional regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Barredo, Principal Investigator — Providence VA Medical Center, Providence, RI
Locations (1):
- Providence VA Medical Center, Providence, RI, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No